CLINICAL TRIAL: NCT04907136
Title: Developing and Testing Health Warning Labels on the ENDS Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: University of Miami (Other)
Responsible Party: Principal Investigator, Wasim Maziak, MD, PhD, Professor, Department of Epidemiology, Florida International University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R01DA051836 (NIH)
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Electronic Cigarette Use
Keywords: Health Warning Labels
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: During this research project, HWLs will be tested on the ENDS device in a clinical lab cross-over study, where each subject uses ENDS in 2 sessions; 1) their preferred product without HWL (control), and 2) their preferred product with pictorial HWL on the ENDS device. This design will test the main study hypothesis: compared to control, using ENDS with the HWLs is associated with decreased satisfaction, dependence suppression, and puffing behavior, but increased knowledge about harm and intention to quit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preferred ENDS (Experimental): All participants will complete a lab visit where they will use their preferred ENDS ad libitum for up to 60 minutes
  Interventions: Other: Preferred ENDS; Other: Preferred ENDS with HWL
- Preferred ENDS with HWL (Experimental): All participants will complete a lab visit where they will use their preferred ENDS with a HWL on the device ad libitum for up to 60 minutes
  Interventions: Other: Preferred ENDS; Other: Preferred ENDS with HWL

INTERVENTIONS:
Other: Preferred ENDS — Preferred ENDS without HWL on device
Other: Preferred ENDS with HWL — Preferred ENDS with a HWL on device

SUMMARY:
In this project, after systematically developing electronic nicotine delivery systems (ENDS) pictorial health warning labels (HWLs), a proven clinical lab model will be used to examine and test their effect when these are placed on the ENDS device on a variety of subjective (e.g. satisfaction, harm perception, nicotine dependence, intention to quit) and objective outcomes (e.g. plasma nicotine, puff topography) in young adults.

DETAILED DESCRIPTION:
The use of electronic nicotine delivery systems (ENDS or e-cigarettes) has reached epidemic levels among young people in the United States (US). ENDS emit toxic substances, including nicotine that irreversibly affects youth's developing brain leading to dependence and increased risk of cigarette smoking initiation, yet misperceptions about their safety are widespread. Therefore, health communication of ENDS-related risks through Health Warning Labels (HWLs) has been considered as a priority by leading health and regulatory bodies in the US to reduce ENDS use among young people. The FIU Epidemiology Clinical Tobacco Research Lab has developed and pilot-tested a clinical lab model to examine the potential effects of pictorial HWLs on young (21-29 yrs) ENDS users' experiences. In this proposal, this model, coupled with a systematic development of ENDS pictorial HWLs, will be used to test their effect when they are placed on the device on a variety of subjective (e.g. satisfaction, harm perception, nicotine dependence, intention to quit) and objective outcomes (e.g. plasma nicotine, puff topography). This will be done in three stages. First, the literature will be reviewed to develop candidate messages and their associated pictures for the HWLs. This initial set of HWLs will then be revised and ranked through a Delphi study among tobacco control, regulation, and health communication experts. Second, focus groups with young ENDS (21-29 yrs) users will be conducted to adapt the candidate HWLs to our target population and device itself. Third, HWLs on the ENDS device will be tested in a clinical lab cross-over study, where each subject uses ENDS in 2 sessions; 1) their preferred product without HWL (control), and 2) their preferred product with pictorial HWL on the ENDS device. This design will test our main hypothesis; compared to control, using ENDS with the HWLs is associated with decreased satisfaction, dependence suppression, and puffing behavior, but increased knowledge about harm and intention to quit. This project will guide policymakers into the application of effective HWLs for ENDS and will develop warning messages and pictorials that national and state stakeholders can use through different modalities in counter-marketing campaigns to protect young people and discourage harmful ENDS use.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy individuals (determined by physical examination).
* Age of 21-35 years.
* Is willing to provide informed consent.
* Is willing to attend the lab as required by the study protocol.
* ENDS users (defined as using ENDS either daily or occasionally in the past 30 days)
* Have abstained from ENDS use for 12 hours prior to each session.

Exclusion Criteria:

* Report smoking cigarettes regularly (> 5 cigarettes/month in the past year).
* Report regular use of any other tobacco/nicotine product (e.g., e-cig, pipes, cigars) in the past year.
* Women who are breast-feeding or test positive for pregnancy (by urinalysis at screening).
* Individuals with self-reported history of chronic disease or psychiatric conditions.
* Individuals with history of or active cardiovascular disease, low or high blood pressure, seizures, and regular use of prescription medications (other than vitamins or birth control).
* Individuals that report current THC (marijuana) smoking/vaping.
* Individuals that report the use of non-commercial (i.e., street) e-cigarette liquid or products
* Individuals that report current EVALI or COVID-19 related symptoms (i.e., cough, shortness of breath, chest pain, nausea, vomiting, abdominal pain, diarrhea, fever, chills, or weight loss)
* Individuals that have or have been exposed to COVID-19 in the last 14 days.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Plasma nicotine | During the 2 participant visits. Blood will be taken 2 times in each ENDS use session: before and after an approximately 60-min ad lib use period
  Change in plasma nicotine level

SECONDARY OUTCOMES:
Puff topography | Time Frame: During participants' two study visits. Puffing behavior is continuously measured during each ENDS use session (an approximately 60-min ad lib use period)
  Measurement of puffing behavior
Minnesota Nicotine Withdrawal Scale | During participants' 2 study visits. Questionnaire will be administered 2 times in each ENDS use session: before and after an approximately 60-min ad lib use period
  This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 11 items scored 0 - 100. These items are presented as Visual Analog Scale with item (measure) centered above a horizontal line anchored on the left with not at all and on the right with extremely.
Tiffany-Drobes Questionnaire of Smoking Urges | During participants' two study visits. Questionnaire will be administered 2 times in each ENDS use session: before and after an approximately 60-min ad lib use period.
  This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 10 items that are scored 0 - 7. Rated on a 7-point Likert scale ranging from 0 (strongly disagree) to 6 (strongly agree).
Carbon monoxide levels | During participants' two study visits. Carbon monoxide levels will be measured 2 times in each ENDS use session: before and after an approximately 60-min ad lib use period
  Change in carbon monoxide levels (in parts per million)
Harm perception | During participants' two study visits. Questionnaire will be administered after each of the 2 ENDS use sessions. Each session is approximately 60-min ad lib use period.
  This scale will assess waterpipe harm perception and measure perceptions of waterpipe relative risk compared to cigarettes. The scale will be scored on a 7-point scale ranging from 1 (not at all harmful), to 7 (extremely harmful).
Duke Sensory Questionnaire | During participants' two study visits. Questionnaire will be administered after each of the 2 ENDS use sessions. Each session is approximately 60-min ad lib use period.
  This scale will assess participants sensory experience of the inhaled product. The scale has nine items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).
The Cigarette/ENDS Evaluation Scale (WES) | During participants' two study visits. Questionnaire will be administered after each of the 2 ENDS use sessions. Each session is approximately 60-min ad lib use period.
  This scale assesses participants' perception of ENDS use. The scale has 11 items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).
Forced expiratory volume (FEV1) | During participants' 2 study visits. FEV tests will be measured 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  Forced expiratory volume (FEV) measures how much air a person can exhale during a forced breath.FEV is used to measure lung function.
Forced vital capacity (FVC) | During participants' 2 study visits. FVC tests will be measured 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  Forced vital capacity (FVC) is the maximum amount of air that can be exhaled when blowing out as fast as possible FVC is used to measure lung function.
Peak expiratory flow (PEF) | During participants' 2 study visits. PEF tests will be measured 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  Peak expiratory flow (PEF) is the maximal flow that can be exhaled when blowing out at a steady rate. PEF is used to measure lung function.
Forced expiratory flow | During participants' 2 study visits. Forced expiratory flow tests will be measured 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  Forced expiratory flow, also known as mid-expiratory flow; the rates at 25%, 50% and 75% FVC are given. Forced expiratory flowis used to measure lung function.

OTHER OUTCOMES:
Heart rate | During participants' two study visits. Heat rate will be measured from baseline continuously throughout each approximately 60-min session.
  Change in heart rate, measured in beats per minute
Blood pressure | During participants' two study visits. Blood pressure will be measured from baseline continuously throughout each approximately 60-min session
  Change in blood pressure, measured in mm/hg

CONTACTS AND LOCATIONS:
Overall Officials: Wasim Maziak, MD, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No